CLINICAL TRIAL: NCT00719810
Title: A Randomized, Double-Blind, Multicenter Study of the Safety and Efficacy of RX 3341 Compared With Tigecycline for the Treatment of Complicated Skin and Skin Structure Infections
Brief Title: Safety and Efficacy Study of a Fluoroquinolone to Treat Complicated Skin Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RX-3341-201
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Results first posted 2010-02-03 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-06

CONDITIONS: Skin Structure Infections; Bacterial Skin Diseases; Staphylococcal Skin Infections
Keywords: complicated; skin
MeSH Terms: conditions — Skin Diseases, Bacterial; Staphylococcal Skin Infections | interventions — delafloxacin; Tigecycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: delafloxacin
- 2 (Experimental)
  Interventions: Drug: delafloxacin
- 3 (Active Comparator)
  Interventions: Drug: tigecycline

INTERVENTIONS:
Drug: delafloxacin — 300 mg intravenous every 12 hours
  Arms: 1
Drug: delafloxacin — 450 mg intravenous every 12 hours
  Arms: 2
Drug: tigecycline — 100 mg then 50 mg intravenous tigecycline every 12 hours
  Arms: 3

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of RX-3341 (delafloxacin), a fluoroquinolone, versus tigecycline, a glycylcycline antibacterial drug, in the treatment of complicated skin and skin structure infections.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years of age) men or women with cSSSI
* Diagnosis of one of the following 3 types of cSSSI: wound infection that has developed within 30 days of surgery, trauma, or a bite injury; abscess that has developed in the 7 days before enrollment; or cellulitis that has developed in the 7 days before enrollment
* Sexually active men and women of childbearing potential must agree to use an acceptable form of contraception, as determined by the investigator, during participation in the study and for 30 days after the final dose of study drug
* The patient must be willing to comply with protocol requirements

Exclusion Criteria:

* Medical history of hypersensitivity or allergic reaction to quinolones, tetracycline or tetracycline derivatives
* Chronic or underlying skin condition at the site of infection
* Infection involving prosthetic materials or foreign bodies (unless prosthetic material will be removed within 24 hours), infection associated with a human bite, osteomyelitis, decubitus ulcer, diabetic foot ulcer, septic arthritis, mediastinitis, necrotizing fasciitis, myositis, tendinitis, endocarditis, toxic shock syndrome, gangrene or gas gangrene, burns covering ≥10% of body surface area, severely impaired arterial blood supply, current evidence of deep vein thrombosis or superficial thrombophlebitis
* An infection that would normally have a high cure rate after surgical incision alone
* Any infection expected to require other antimicrobial agents in addition to study drug
* Receipt of >24 hours of systemic antibiotic therapy in the 7 days before enrollment
* A severely compromised immune system
* History of Child-Pugh Class B or C liver disease or severe renal impairment (creatinine clearance of <30 mL/minute)
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Breen, MD, Study Director — Melinta Therapeutics, Inc.
Locations (14):
- United States (13):
  - Physician Alliance Research Center, Anaheim, California
  - Quality of Life Medical Center, LLC, Hawaiian Gardens, California
  - Tri City Medical Center, Oceanside, California
  - Crest Clinical Trials, Santa Ana, California
  - Internal Medicine Associates of Lee County, Fort Myers, Florida
  - Joseph M. Still Research Foundation, Inc., Augusta, Georgia
  - Southeast Regional Research Group, Columbus, Georgia
  - Southeast Regional Research Group, Ludowici, Georgia
  - Southeast Regional Research Group, Savannah, Georgia
  - St. James Health Care, Butte, Montana
  - Riverside Methodist Hospital, Columbus, Ohio
  - West Houston Clinical Research Services, Houston, Texas
  - Westbury Medical Clinic, Houston, Texas
- Clinical Research Puerto Rico, Inc, San Juan, Puerto Rico

REFERENCES:
- [Derived] O'Riordan W, Mehra P, Manos P, Kingsley J, Lawrence L, Cammarata S. A randomized phase 2 study comparing two doses of delafloxacin with tigecycline in adults with complicated skin and skin-structure infections. Int J Infect Dis. 2015 Jan;30:67-73. doi: 10.1016/j.ijid.2014.10.009. Epub 2014 Oct 30. PMID 25448332

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study targeted participants with complicated skin and skin structure infections (cSSSI), i.e. infections involving subcutaneous tissues or requiring surgical intervention. Patients could have one of three infection types: wound infection, abscess, or cellulitis.
Period: Overall Study
Arm/Group | Delafloxacin 300 mg IV q12h | Delafloxacin 450 mg IV q12h | Tigecycline 100 mg IV x 1, Followed by 50 mg IV q12h
Started | 49 | 51 | 50
Completed | 46 | 47 | 42
Not Completed | 3 | 4 | 8
Not completed — Adverse Event | 0 | 2 | 3
Not completed — Lost to Follow-up | 2 | 0 | 3
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delafloxacin 300 mg IV q12h | Delafloxacin 450 mg IV q12h | Tigecycline 100 mg IV x 1, Followed by 50 mg IV q12h | Total
Number analyzed (Participants) | 49 | 51 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (15.10) | 37.2 (14.35) | 40.4 (13.83) | 40.1 (14.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 15 | 48
  Male | 31 | 36 | 35 | 102

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response at Test of Cure (TOC) in the Clinically Evaluable (CE) Population
Description: A Cure was defined as resolution of baseline signs and symptoms, or improvement to an extent that no additional antibiotic treatment is necessary. Failure was defined as the need for additional antibiotics, either because of lack of efficacy after at least 2 days (i.e., 4 doses) of study treatment or because of treatment-related adverse events (AEs), and/or the need for surgical intervention greater than 48 hours after study entry.
Time Frame: 14-21 days after the last dose of study drug
Population: The CE population included patients with a diagnosis of cSSSI who received at least 80% of study drug, had a test of cure (TOC) visit 14-21 days after the last dose of study drug, and who did not receive any concomitant, systemic antibacterial therapy with activity against the causative pathogen.
Measure: Number; unit: Participants
Arm/Group | Delafloxacin 300 mg IV q12h | Delafloxacin 450 mg IV q12h | Tigecycline 100 mg IV x 1, Followed by 50 mg IV q12h
Number analyzed (Participants) | 35 | 40 | 34
Participants | 33 | 37 | 31

2. Secondary Outcome: Clinical Response in Patients With Methicillin-resistant Staphylococcus Aureus (MRSA)
Description: as for outcome 1
Time Frame: 14-21 days after the last dose of study drug
Population: Clinically Evaluable (CE) patients (see previous definition) with MRSA isolated from screening culture of primary infection.
Measure: Number; unit: Participants
Arm/Group | Delafloxacin 300 mg IV q12h | Delafloxacin 450 mg IV q12h | Tigecycline 100 mg IV x 1, Followed by 50 mg IV q12h
Number analyzed (Participants) | 14 | 20 | 14
Participants | 13 | 19 | 12

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) that occurred from the time the patient signed the informed consent form (ICF) were to be reported on the appropriate electronic case report form (eCRF).
Arm/Group | Delafloxacin 300 mg IV q12h | Delafloxacin 450 mg IV q12h | Tigecycline 100 mg IV x 1, Followed by 50 mg IV q12h
Serious Adverse Events (participants affected / at risk) | 1/49 | 3/51 | 3/50
Other Adverse Events (participants affected / at risk) | 14/49 | 32/51 | 36/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delafloxacin 300 mg IV q12h (N=49) | Delafloxacin 450 mg IV q12h (N=51) | Tigecycline 100 mg IV x 1, Followed by 50 mg IV q12h (N=50)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delafloxacin 300 mg IV q12h (N=49) | Delafloxacin 450 mg IV q12h (N=51) | Tigecycline 100 mg IV x 1, Followed by 50 mg IV q12h (N=50)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 12 (12) | 5 (5)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4)
Fatigue (General disorders) | 0 (0) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 4 (4) | 6 (6)
Infusion site pain (General disorders) | 0 (0) | 7 (7) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 13 (13) | 23 (23)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (3)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 6 (6) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor retains control of all publication rights.